CLINICAL TRIAL: NCT03985787
Title: The Effects of Resistance Training on Appetite Regulation
Brief Title: Resistance Training and Appetite Regulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 18-1298; 1R21DK115200-01A1 (NIH)
Record Dates: First submitted 2019-04-11; First posted 2019-06-14 (Actual); Last update posted 2021-09-28 (Actual); Status verified 2021-09

CONDITIONS: Obesity
Keywords: Resistance Exercise; Appetite Regulation
MeSH Terms: conditions — Obesity | interventions — Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All Participants (Experimental): 12-weeks of a full body resistance training intervention. Intervention will consist of 4 training sessions per week that are approximately 45-minutes in length. Two days will be upper body training and 2 days lower body
  Interventions: Behavioral: Resistance Training

INTERVENTIONS:
Behavioral: Resistance Training — 12-weeks of a full body resistance training intervention. Intervention will consist of 4 training sessions per week that are approximately 45-minutes in length. Two days will be upper body training and 2 days lower body

SUMMARY:
This study plans to learn more about how resistance training impacts appetite and the brain's response to food. The study will be evaluating how the brain responds to food images as well as how behaviors and hormones change with a 12 week resistance training intervention.

DETAILED DESCRIPTION:
Aim 1: To determine if RT impacts neuronal function associated with food intake behavior in a manner favoring reduced EI in overweight/obese adults.

Hypothesis: Compared to pre, post-RT fMRI measures will demonstrate ↓ neuronal responses to food cues in the insula, prefrontal cortex, and hypothalamus, brain regions implicated in reward, impulsivity, motivation, and regulation of ingestive behaviors. These changes will be associated with ad libitum EI.

Aim 2: To determine if RT impacts appetite-related peptides, ratings, and food intake behaviors in a manner favoring reduced EI in overweight/obese adults.

Hypothesis: Compared to pre, post-RT measures will show changes in appetite-related peptides, ratings (↓ hunger ↑ satiety), and behaviors (↓food-related cravings & impulsivity, ↑ self-efficacy) consistent with EI reduction. Changes in appetite regulation indices will be associated with changes in relevant brain networks (Aim 1). These changes will also be associated with ↓ ad libitum EI.

Exploratory Aim: To determine if RT impacts neuronal function and appetite-related peptides and behaviors in a manner favoring ↓ EI in Non-Compensators (top tertile of fat mass loss) as compared to Compensators (bottom tertile of fat mass loss).

Hypothesis: Compared to Compensators, Non-Compensators will show ↓ neuronal responses to food cues and default network, and changes in appetite-related peptides, ratings, and behaviors consistent with ↓ EI.

ELIGIBILITY:
Inclusion Criteria:

* all ethnic groups
* both sexes
* age: 18-55
* BMI: 27-40 kg/m2
* weight stable (±5% in last 6 months)
* sedentary (<2 hours of planned physical activity/week by self-report, no RT in previous 12-months)

Exclusion Criteria:

* history of CVD
* DM
* uncontrolled Hypertension
* untreated thyroid disease
* renal disease
* hepatic disease
* other condition affecting weight/metabolism
* unable to exercise
* smoker
* medications affecting weight
* EI or EE in past 6 months
* weight loss/gain >5% in past 6 months
* post-menopausal women (defined as age appropriate women with 6 months or more of amenorrhea)
* currently pregnant, lactating, < 6 months post-partum
* woman who have undergone oophorectomy
* bariatric surgery
* major psychiatric disorder
* alcohol or substance abuse
* depression by history and/or score >21 on CES-D
* history of eating disorders and/or score >20 on EATS-26

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2018-10-24 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2021-05-31 (Actual)

PRIMARY OUTCOMES:
Change in Neuronal Responses to Food Cues in Regions of Interest | Baseline, 12 Weeks
  Changes in the insula, prefrontal cortex, and hypothalamus response to salient food cues (pre vs post-RT) as measured by fMRI in response to 12-weeks of RT

SECONDARY OUTCOMES:
Change in Whole Brain Response | Baseline, 12 Weeks
  Whole brain changes in response to salient food cues (pre vs post RT) as measured by fMRI in response to 12-weeks of RT
Change in Default Mode Network | Baseline, 12 Weeks
  Changes in the DMN resting state activity and large-scale network connectivity (pre vs post RT) as measured by MRI in response to 12-weeks of RT
Changes in Appetite Ratings | Baseline, 12 Weeks
  Changes in measures of appetite (hunger, satiety, and prospective food consumption) area under the curve [AUC] following a standardized test-meal in response to 12-weeks of RT.
Changes in Appetite-Related Hormones | Baseline, 12 Weeks
  Changes in appetite-related hormones [ghrelin, PYY, and GLP-1] area under the curve [AUC] following a standardized test meal in response to 12-weeks of RT.
Change in In Lab Ad Libitum Energy Intake (kcals) | Baseline, 12 Weeks
  Change in In lab ad libitum buffet lunch (via weigh and measure methodology) three hours after breakfast test meal at baseline and post-intervention
Change in Free-Living Ad libitum Energy Intake (kcals) | Baseline, 12 Weeks
  Change in Three days of free-living ad libitum energy intake (via DHQ food frequency questionnaire) at baseline and post intervention.

OTHER OUTCOMES:
Changes in Free-Living Physical Activity and Sedentary Time | Baseline, 12 Weeks
  Physical Activity and Sedentary Time will be measured via activPAL (PALTechnologies: Glasgow, Scotland) activity monitor. Participants will be instructed to wear the monitor on their right leg for 7 consecutive days at all times except when sleeping or participating in water-based activities (e.g. showering, swimming). The time-stamped "event" data file from the activPAL software will be used to determine time spent sitting/lying, standing and stepping per day.
Changes in Muscular Strength | Baseline, 12 Weeks
  Muscular Strength via 10 repetition maximum of chest and leg press on strength training machines, respectively.
Change in Body Mass (kg) | Baseline, 12 Weeks
  Via Digital scale
Change in Body Composition | Baseline, 12 Weeks
  Assessment of fat mass and lean mass via DXA scan
Change in Neuronal Responses to Food Cues in Regions of Interest by Non-Compensator vs. Compensator groups | Baseline, 12 Weeks
  Changes in the insula, prefrontal cortex, and hypothalamus response to salient food cues (pre vs post-RT) as measured by fMRI in response to 12-weeks of RT. "Non-Compensators" (will be defined as those who lose weight in response to the 12-week resistance training intervention. "Compensators" will be defined as those who maintain or gain weight in response to the 12-week resistance training interventions.
Change in Neuronal Responses to Food Cues in Regions of Interest by Sex | Baseline, 12 Weeks
  Changes in the insula, prefrontal cortex, and hypothalamus response to salient food cues (pre vs post-RT) as measured by fMRI in response to 12-weeks of RT.
Change in Whole Brain Response by Non-Compensator vs. Compensator groups | Baseline, 12 Weeks
  Whole brain changes in response to salient food cues (pre vs post RT) as measured by fMRI in response to 12-weeks of RT. "Non-Compensators" (will be defined as those who lose weight in response to the 12-week resistance training intervention. "Compensators" will be defined as those who maintain or gain weight in response to the 12-week resistance training interventions.
Change in Whole Brain Response by Sex | Baseline, 12 Weeks
  Whole brain changes in response to salient food cues (pre vs post RT) as measured by fMRI in response to 12-weeks of RT.
Change in Default Mode Network by Non-Compensator vs. Compensator groups | Baseline, 12 Weeks
  Changes in the DMN resting state activity and large-scale network connectivity (pre vs post RT) as measured by MRI in response to 12-weeks of RT. "Non-Compensators" (will be defined as those who lose weight in response to the 12-week resistance training intervention. "Compensators" will be defined as those who maintain or gain weight in response to the 12-week resistance training interventions.
Change in Default Mode Network by Sex | Baseline, 12 Weeks
  Changes in the DMN resting state activity and large-scale network connectivity (pre vs post RT) as measured by MRI in response to 12-weeks of RT.
Changes in Appetite Ratings by Non-Compensator vs. Compensator groups | Baseline, 12 Weeks
  Changes in measures of appetite (hunger, satiety, and prospective food consumption) area under the curve [AUC] following a standardized test-meal in response to 12-weeks of RT. "Non-Compensators" (will be defined as those who lose weight in response to the 12-week resistance training intervention. "Compensators" will be defined as those who maintain or gain weight in response to the 12-week resistance training interventions.
Changes in Appetite Ratings by Sex | Baseline, 12 Weeks
  Changes in measures of appetite (hunger, satiety, and prospective food consumption) area under the curve [AUC] following a standardized test-meal in response to 12-weeks of RT. "
Changes in Appetite-Related Hormones by Non-Compensator vs. Compensator groups | Baseline, 12 Weeks
  Changes in appetite-related hormones [ghrelin, PYY, and GLP-1] area under the curve [AUC] following a standardized test meal in response to 12-weeks of RT. "Non-Compensators" (will be defined as those who lose weight in response to the 12-week resistance training intervention. "Compensators" will be defined as those who maintain or gain weight in response to the 12-week resistance training interventions.
Changes in Appetite-Related Hormones by Sex | Baseline, 12 Weeks
  Changes in appetite-related hormones [ghrelin, PYY, and GLP-1] area under the curve [AUC] following a standardized test meal in response to 12-weeks of RT.
Change in In Lab Ad Libitum Energy Intake (kcals) by Non-Compensator vs. Compensator groups | Baseline, 12 Weeks
  Change in In lab ad libitum buffet lunch (via weigh and measure methodology) three hours after breakfast test meal at baseline and post-intervention. "Non-Compensators" (will be defined as those who lose weight in response to the 12-week resistance training intervention. "Compensators" will be defined as those who maintain or gain weight in response to the 12-week resistance training interventions.
Change in In Lab Ad Libitum Energy Intake (kcals) by Sex | Baseline, 12 Weeks
  Change in In lab ad libitum buffet lunch (via weigh and measure methodology) three hours after breakfast test meal at baseline and post-intervention.
Change in Free-Living Ad libitum Energy Intake (kcals) by Non-Compensator vs. Compensator groups | Baseline, 12 Weeks
  Change in Three days of free-living ad libitum energy intake (via DHQ food frequency questionnaire) at baseline and post intervention. "Non-Compensators" (will be defined as those who lose weight in response to the 12-week resistance training intervention. "Compensators" will be defined as those who maintain or gain weight in response to the 12-week resistance training interventions.
Change in Free-Living Ad libitum Energy Intake (kcals) by Sex | Baseline, 12 Weeks
  Change in Three days of free-living ad libitum energy intake (via DHQ food frequency questionnaire) at baseline and post intervention.
Changes in Free-Living Physical Activity and Sedentary Time by Non-Compensator vs. Compensator groups | Baseline, 12 Weeks
  Physical Activity and Sedentary Time will be measured via activPAL (PALTechnologies: Glasgow, Scotland) activity monitor. Participants will be instructed to wear the monitor on their right leg for 7 consecutive days at all times except when sleeping or participating in water-based activities (e.g. showering, swimming). The time-stamped "event" data file from the activPAL software will be used to determine time spent sitting/lying, standing and stepping per day. "Non-Compensators" (will be defined as those who lose weight in response to the 12-week resistance training intervention. "Compensators" will be defined as those who maintain or gain weight in response to the 12-week resistance training interventions.
Changes in Free-Living Physical Activity and Sedentary Time by Sex | Baseline, 12 Weeks
  Physical Activity and Sedentary Time will be measured via activPAL (PALTechnologies: Glasgow, Scotland) activity monitor. Participants will be instructed to wear the monitor on their right leg for 7 consecutive days at all times except when sleeping or participating in water-based activities (e.g. showering, swimming). The time-stamped "event" data file from the activPAL software will be used to determine time spent sitting/lying, standing and stepping per day.
Change in Muscular Strength by Non-Compensators vs Compensators | Baseline, 12 Weeks
  Muscular Strength via 10 repetition maximum of chest and leg press on strength training machines, respectively. "Non-Compensators" (will be defined as those who lose weight in response to the 12-week resistance training intervention. "Compensators" will be defined as those who maintain or gain weight in response to the 12-week resistance training interventions.
Change in Muscular Strength by Sex | Baseline, 12 Weeks
  Muscular Strength via 10 repetition maximum of chest and leg press on strength training machines, respectively.
Change in Body Mass by Non-Compensator vs. Compensator groups | Baseline, 12 Weeks
  Via Digital scale. "Non-Compensators" (will be defined as those who lose weight in response to the 12-week resistance training intervention. "Compensators" will be defined as those who maintain or gain weight in response to the 12-week resistance training interventions.
Change in Body Mass by Sex | Baseline, 12 Weeks
  Via Digital scale.
Change in Body Composition by Non-Compensator vs. Compensator groups | Baseline, 12 Weeks
  Assessment of fat mass and lean mass via DXA scan. "Non-Compensators" (will be defined as those who lose weight in response to the 12-week resistance training intervention. "Compensators" will be defined as those who maintain or gain weight in response to the 12-week resistance training interventions.
Change in Body Composition by Sex | Baseline, 12 Weeks
  Assessment of fat mass and lean mass via DXA scan.

CONTACTS AND LOCATIONS:
Overall Officials: Marc-Andre Cornier, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Denver - Anschutz Medical Campus, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No